CLINICAL TRIAL: NCT03932630
Title: Looping Whilst Restricting Carbohydrates (LINEAR) - a Randomised Two-Period Crossover Trial
Brief Title: Looping Whilst Restricting Carbohydrates
Acronym: LINEAR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19 related challenges and restrictions, the project could not be launched as planned. Meanwhile, the current state of research has changed and the initialisation of the project is no longer appropriate. No participants were recurited.
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Lia Bally, Head of Metabolic Science Research Group, Insel Gruppe AG, University Hospital Bern
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LINEAR
Record Dates: First submitted 2019-04-28; First posted 2019-05-01 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Diabetes; Type 1 Diabetes
Keywords: artificial pancreas; hybrid closed-loop; low carbohydrate diet; glucose control
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Diet, Carbohydrate-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study intervention (Experimental)
  Interventions: Other: Low carbohydrate diet
- Control intervention (Active Comparator)
  Interventions: Other: balanced diet

INTERVENTIONS:
Other: Low carbohydrate diet — The study intervention will be an eucaloric low carbohydrate diet (15-20 % of carbohydrates) for 2 weeks.
  Arms: Study intervention
Other: balanced diet — The control intervention will be a energy-matched balanced diet (50 % of carbohydrates) for 2 weeks.
  Arms: Control intervention

SUMMARY:
To investigate the efficacy, safety and utility of hybrid closed-loop glucose control during a low carbohydrate vs. iso-energetic balanced diet in individuals with type 1 diabetes.

DETAILED DESCRIPTION:
Closed-loop systems combining an insulin pump, a glucose sensor and a dosing algorithm that adjusts insulin delivery in a glucose-responsive manner achieve significantly better glucose control than conventional therapy in type 1 diabetes. Achieving satisfactory postprandial glucose control, however, continues to be challenging. The main limitation is the delayed pharmacokinetics and -dynamics of subcutaneously administered insulin with peak actions between 1 and 2 hours. Conversely, glucose levels typically rise within 10minutes following carbohydrate intake. This mismatch largely explains the inability of current closed-loop systems to control postprandial glucose excursions and the increased risk of late postprandial hypoglycaemia in response to both user-derived meal bolus administration and reactive algorithm-driven insulin infusion.

Restricting carbohydrate may therefore significantly improve post-prandial glucose control whilst reducing hypoglycaemia. The efficacy of hybrid closed-loop operation in individuals with type 1 diabetes adhering to a low carbohydrate compared to a iso-caloric balanced diet has not been investigated to date.

ELIGIBILITY:
Inclusion Criteria:

* Female and male subjects aged 18 years or older
* Diabetes mellitus Type 1 as definded by WHO for at least 2 years or C-peptide negative (<100 pmol/L with concomitant blood glucose > 4 mmol/L)
* hybrid-closed-loop Insulin therapy (Minimed 670G) for at least 2 months
* HbA1c <= 9 %
* The subject is willing and capable of adhering to the diet plan.

Exclusion Criteria:

* Physical or psychological condition likely to interfere with the normal conduct of the study and interpretation of the study results as judged by the investigator.
* Excess alcohol consumption (> 3 units/day for men, > 2 units/day for women)
* Pregnancy, planned pregnancy or breast feeding
* Current participation in another clinical trial
* Total daily insulin dose >2 IU/kg/day
* Nephrolithiasis
* Hereditary dyslipidemia
* Liver steatosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of time in target glucose range (3.9 - 10.0 mmol/L) | 2 weeks
  The percentage of time in target glucose range will be assessed using continuous glucose monitoring (CGM).

SECONDARY OUTCOMES:
Percentage of time above target (>10 mmol/L) | 2 weeks
  The percentage of time below target (>10 mmol/L) will be assessed using continuous glucose monitoring (CGM).
Percentage of time below target (<3.9 mmol/L) | 2 weeks
  The percentage of time below target (<3.9 mmol/L) will be assessed using continuous glucose monitoring (CGM).
Percentage of time in hypoglycemia (<3.0 mmol/L) | 2 weeks
  The percentage of time in hypoglycemia (<3.0 mmol/L) will be assessed using continuous glucose monitoring (CGM).
Hypoglycemia burden quantified as the area under the curve (AUC) with glucose < 3 mmol/L | 2 weeks
  Hypoglycemia burden will be assessed using continuous glucose monitoring (CGM).
Percentage of time in hyperglycemia (>16.7 mmol/L) | 2 weeks
  The percentage of time in hyperglycemia (>16.7 mmol/L) will be assessed using continuous glucose monitoring (CGM).
Mean glucose levels (mmol/l) | 2 weeks
  Mean sensor glucose levels will be assessed using continuous glucose monitoring (CGM).
Total daily insulin dose (U) | 2 weeks
  Total daily insulin dose will be recorded by the insulin pump
Daily manual bolus Insulin dose (U) | 2 weeks
  Daily manual bolus insulin dose will be recorded by the insulin pump
2 hour postprandial glucose increment (mmol/) | 2 weeks
  2 hour postprandial glucose increment will be assessed using continuous glucose monitoring (CGM).
Within-day standard deviation of glucose (mmol/l) | 2 weeks
  Within-day standard deviation of glucose will be assessed using continuous glucose monitoring (CGM).
Within day coefficient of variation of glucose (%) | 2 weeks
  Within day coefficient of variation of glucose will be assessed using continuous glucose monitoring (CGM).
Between days coefficient of variation of glucose (%) | 2 weeks
  Between days coefficient of variation of glucose will be assessed using continuous glucose monitoring (CGM).
Night-time percentage of time in target glucose range (3.9 - 10.0 mmol/L) | Between 00:00-06:00 over 2 weeks
  Percentage of time in target glucose range will be assessed using continuous glucose monitoring (CGM).
Night-time percentage of time above target (> 10.0 mmol/L) | Between 00:00-06:00 over 2 weeks
  Percentage of time above target will be assessed using continuous glucose monitoring (CGM).
Night-time percentage of time below target (< 3.9 mmol/L) | Between 00:00-06:00 over 2 weeks
  Percentage of time below target will be assessed using continuous glucose monitoring (CGM).
Night-time percentage of time in hypoglycemia (< 3.0 mmol/L) | Between 00:00-06:00 over 2 weeks
  Percentage of time in hypoglycemia will be assessed using continuous glucose monitoring (CGM).
Night-time percentage of time in hyperglycemia (> 16.7 mmol/L) | Between 00:00-06:00 over 2 weeks
  Percentage of time in hyperglycemia will be assessed using continuous glucose monitoring (CGM).
Night-time mean glucose levels | Between 00:00-06:00 over 2 weeks
  Mean sensor glucose levels will be assessed using continuous glucose monitoring (CGM).
Within night-time standard deviation of glucose (mmol/l)compared to within daytime period (06: - 24:00) standard deviation of glucose (mmol/l) | Between 00:00-06:00 over 2 weeks
  Standard deviation of glucose will be assessed using continuous glucose monitoring (CGM).
Within nighttime coefficient of variation of glucose(%) | Between 00:00-06:00 over 2 weeks
  Coefficient of variation of glucose (%) will be assessed using continuous glucose monitoring (CGM).
Change from baseline in lipid profile | 2 weeks
  Plasma Lipid profile (total Cholesterol, LDL-Cholesterol, HDL-Cholesterol, Triglycerides)
Total daily calorie intake (kcal/day) | 2 weeks
  Total daily calorie intake will be assessed based on photo-documentation of dietary intake
Mean beta-hydroxy butyrate level | 2 weeks
  based on download of blood Ketone meter
Change from baseline in fasting plasma metabolome | 2 weeks
  Fasting serum sampling
Incidence of (serious) adverse events | 12 weeks
  Incidence of severe hypoglycaemia, signficant hyperglycaemia with ketonemia, other SAEs, adverse events, adverse defice effects and device deficiencies
Percentage of time when pump was in Auto-mode | 2 weeks
  Based on pump data download

CONTACTS AND LOCATIONS:
Overall Officials: Lia Bally, MD PhD, Principal Investigator — Inselspital, Bern University Hospital, University of Bern
Locations (1):
- University Department of Endocrinology, Diabetology, Clinical Nutrition and Metabolism, Bern, Switzerland